CLINICAL TRIAL: NCT00141076
Title: Glycemic Index, Obesity, Insulin Resistance and CVD Risk, Part 2
Brief Title: Glycemic Index and CVD: a Crossover Feeding Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Charles H. Hood Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 59240-#2; R01DK059240 (NIH); 2002-P-001495/22 (BWH)
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Obesity
Keywords: obesity; glycemic index; insulin resistance; cardiovascular disease; diabetes
MeSH Terms: conditions — Obesity; Insulin Resistance; Cardiovascular Diseases; Diabetes Mellitus

INTERVENTIONS:
Behavioral: low vs high glycemic index diet

SUMMARY:
This study will compare the physiological effects of two isoenergetic, nutrient-controlled diets that differ in glycemic index. The diets will be studied in obese adults in a 10-day crossover feeding trial.

DETAILED DESCRIPTION:
This study will compare the physiological effects of two isoenergetic, nutrient-controlled diets that differ in glycemic index. The diets will be studied in obese male adults in a 10-day crossover feeding trial. Hypothesis: Obese subjects will show improvements in clinical endpoints associated with risk for diabetes and cardiovascular disease (CVD) after consuming a controlled low (compared to high) glycemic index diet for 10 days. 1º endpoint: insulin sensitivity as measured by the modified Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT). 2º endpoints: CVD risk factors; postprandial studies of oxidative stress; thermic effect of food.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 35 years
* male
* BMI ≥ 27 ≤45 kg/m2
* willingness to refrain from alcohol and caffeinated beverage consumption for duration of study

Exclusion Criteria:

* major medical illness
* an abnormal screening laboratory test
* taking any prescription medications that might affect body weight
* current smoking (1 cigarette during any of the last 7 days)
* consuming special diets

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2003-10; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity as measured by FS-IVGTT

SECONDARY OUTCOMES:
CVD risk factors
Postprandial studies of oxidative stress
Thermic effect of food

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Diego Botero, MD, Study Director — Boston Children's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States